CLINICAL TRIAL: NCT05261139
Title: A PHASE 2/3, INTERVENTIONAL SAFETY, PHARMACOKINETICS, AND EFFICACY, OPEN-LABEL, MULTI-CENTER, SINGLE-ARM STUDY TO INVESTIGATE ORALLY ADMINISTERED PF-07321332 (NIRMATRELVIR)/RITONAVIR IN NONHOSPITALIZED SYMPTOMATIC PEDIATRIC PARTICIPANTS WITH COVID-19 WHO ARE AT RISK OF PROGRESSION TO SEVERE DISEASE
Brief Title: EPIC-Peds: A Study to Learn About the Study Medicine Called PF-07321332 (Nirmatrelvir)/Ritonavir in Patients Under 18 Years of Age With COVID-19 That Are Not Hospitalized But Are at Risk for Severe Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C4671026; 2023-509773-23-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-02-25; First posted 2022-03-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: Severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2); Pediatrics
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Cohort 1 nirmatrelvir/ritonavir (Experimental): nirmatrelvir/ritonavir will be given by tablets or powder by mouth twice a day for 5 days (10 doses total).
  Weight ≥40 kg
  1. ≥12 to <18 years
  2. ≥6 to <12 years
  Interventions: Drug: nirmatrelvir; Drug: ritonavir
- Cohort 2 nirmatrelvir/ritonavir (Experimental): nirmatrelvir/ritonavir will be given as powder by mouth twice a day for 5 days (10 doses total) Weight ≥20 to <40 kg, ≥6 to <18 years
  Interventions: Drug: nirmatrelvir; Drug: ritonavir
- Cohort 3 nirmatrelvir/ritonavir (Experimental): nirmatrelvir/ritonavir
  ≥2 to <6 years
  Interventions: Drug: nirmatrelvir; Drug: ritonavir
- Cohort 4 nirmatrelvir/ritonavir (Experimental): nirmatrelvir/ritonavir
  ≥1 month (≥28 days) to <2 years
  Interventions: Drug: nirmatrelvir; Drug: ritonavir
- Cohort 5 nirmatrelvir/ritonavir (Experimental): nirmatrelvir/ritonavir <1 month (<28 days) old
  Interventions: Drug: nirmatrelvir; Drug: ritonavir

INTERVENTIONS:
Drug: nirmatrelvir — PF-07321332
Drug: ritonavir — ritonavir

SUMMARY:
The purpose of this clinical trial is to learn about the safety, pharmacokinetics (pharmacokinetics helps us understand how the drug is changed and eliminated from your body after you take it), and efficacy (how well a study treatment works in the study) of the study medicine (called nirmatrelvir/ritonavir) for potential treatment of coronavirus disease 2019 (COVID-19).

The study medicine will be given to patients under 18 years of age with COVID-19 that are not hospitalized but are at risk for severe disease.

ELIGIBILITY:
Inclusion criteria:

* Male and female, age 0 to < 18 years, able to swallow for some participants
* Confirmed SARS-CoV-2 infection within 72 hours prior to enrollment
* Initial onset of COVID-19 signs/symptoms within 5 days prior to the day of enrollment and at least 1 of the specified COVID-19 signs/symptoms present at enrollment
* Has at least 1 characteristic or underlying medical condition associated with an increased risk of developing severe illness from COVID-19

Exclusion Criteria:

* History of or need for hospitalization for the medical treatment of COVID-19
* Total bilirubin >=2X upper limit of normal (ULN) (except for Gilbert's syndrome)
* Receiving dialysis or have known moderate to severe renal impairment
* Suspected or confirmed concurrent active systemic infection other than COVID-19
* History of hypersensitivity or other contraindication to any of the components of the study intervention
* Current or expected use of any medications or substances that are highly dependent on CYP3A4 for clearance or strong inducers of cytochrome P450 (CYP)3A4
* Has received or is expected to receive antibody treatment, antiviral treatment or convalescent COVID-19 plasma
* Participating in another interventional clinical study with an investigational compound or device, including those for COVID-19 through the study follow up
* Females who are pregnant or breastfeeding

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Cohort 1-2: Maximum Observed Plasma Concentration (Cmax) of nirmatrelvir and ritonavir | Day 1: 1 hour-post dose; Day 4: pre-dose; Day 5: pre-dose, and 1, and 2 hours post dose
Cohort 1-2: Area Under the Curve to the End of the Dosing Period (AUC0-tau) of nirmatrelvir and ritonavir | Day 1: 1 hour-post dose; Day 4: pre-dose; Day 5: pre-dose, and 1, and 2 hours post dose
Incidence of Treatment Emergent Adverse Events (TEAEs) leading to discontinuations. | From Baseline up through Day 34
Incidence of Serious Adverse Events (SAEs) leading to discontinuations. | From Baseline up through Day 34
Incidence of Adverse Events (AEs) leading to discontinuations. | From Baseline up through Day 34
Number of participants with change from Baseline in Vital Signs | From Baseline up through Day 34

SECONDARY OUTCOMES:
Viral load assessment titers measured via reverse transcription polymerase chain reaction (RT-PCR) in nasopharyngeal or nasal swabs over time | Baseline, Day 5, 6, 10, 14 and 28
Proportion of participants with COVID-19 related hospitalization or death from any cause | From Baseline through Day 28
Patient assessment on acceptability and palatability of nirmatrelvir/ritonavir (film-coated tablets and oral powder) | At baseline only for tablets and after each dose for powder formulation
  Frequency of responses to visual questionnaire on taste.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (73):
- United States (50):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente, Los Angeles, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - UCLA, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Life Spring Research Foundation, Miami, Florida
  - Children's Healthcare of Atlanta - Arthur M. Blank Hospital, Atlanta, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Louisiana State University Health Sciences Shreveport, Shreveport, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Childrens Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - St. Louis Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - University of New Mexico Hospital, COVID-19 Research Clinic, Albuquerque, New Mexico
  - University of New Mexico Clinical and Translational Science Center, Albuquerque, New Mexico
  - Suny University at Buffalo, Buffalo, New York
  - Advanced Specialty Care, Commack, New York
  - Stony Brook Medicine Clinical Research Center, East Setauket, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Columbia University Irving Medical Center, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Upstate Health Care Center, Syracuse, New York
  - Crouse Physicians Office Building, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Upstate Golisano Children's Hospital, Syracuse, New York
  - Clinical and Translational Research Center, Chapel Hill, North Carolina
  - investigational Drug Services Pharmacy, UNC Hospitals, Chapel Hill, North Carolina
  - UNC Children's Hospital, Chapel Hill, North Carolina
  - UNC Global Clinical Research North, Chapel Hill, North Carolina
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - UNC Children's Raleigh, Raleigh, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - UH Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Parma Medical Center, Parma, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital-Clinical Trials, Providence, Rhode Island
  - Avera McKennan Hospital & University Health Center, Sioux Falls, South Dakota
  - Avera Research Institute - Sioux Falls, Sioux Falls, South Dakota
  - Texas Children's Hospital, Houston, Texas
  - Biopharma Informatic, LLC, McAllen, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - University of Utah, Salt Lake City, Utah
- Bulgaria (5):
  - МHAT "Sveti Ivan Rilski" Gorna Oryahovitsa, Gorna Oryahovitsa
  - "Specialized Hospital for Active Treatment of Pneumo-Physiatric Diseases Dr. Dimitar Gramatikov -, Rousse
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - DCC "Alexandrovska", Sofia
  - Specialized Hospital for Active Treatment of Pneumo-Phthisiatric Diseases Vratsa EOOD, Vratsa
- Japan (2):
  - Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo
  - Osaka City General Hospital, Osaka
- Mexico (11):
  - Instituto Nacional de Pediatria, Mexico City, Mexico City
  - Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico City
  - JM Research SC, Cuernavaca, Morelos
  - Fundación Santos y De la Garza Evia, Monterrey, Nuevo León
  - Eukarya Pharmasite S.C., Monterrey, Nuevo León
  - Unidad de Atención Médica e Investigación en Salud, Mérida, Yucatán
  - Kohler & Milstein Research S.A. De C.V., Mérida, Yucatán
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatán S., Mérida, Yucatán
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Arké SMO S.A de C.V, Veracruz
  - Sociedad de Metabolismo y Corazon S.C., Veracruz
- San Miguel Medical, Trujillo Alto, Puerto Rico
- South Africa (3):
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - CRISMO Research Centre, Germiston, Gauteng
  - Botho Ke Bontle Health Services, Pretoria, Gauteng
- St. George's Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671026